CLINICAL TRIAL: NCT05097118
Title: Surgical Site Infiltration Using Ketamine Versus Bupivacaine for Analgesia in Post-operative Appendectomy Operation
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Gehad Ahmed Aly, resident doctor at Anaesthesia and ICU department sohag university hospital, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-21-10-03
Record Dates: First submitted 2021-10-17; First posted 2021-10-27 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Appendicitis Acute
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group of Ketamine injection (Experimental): Ketamine infiltration for post operative analgesia
  Interventions: Drug: Ketamine Versus Bupivacaine
- Group of Bupivacaine injection (Experimental): Bupivacaine infiltration for post operative analgesia
  Interventions: Drug: Ketamine Versus Bupivacaine

INTERVENTIONS:
Drug: Ketamine Versus Bupivacaine — Drugs Ketamine versus Bupivacaine

SUMMARY:
surgical site infiltration using ketamine versus Bupivacaine for analgesia in post-operative Appendectomy operation by Ketamine versus Bupivacaine

ELIGIBILITY:
Inclusion Criteria:

* 60 adult patients with ASA physical physical status class 1 and class 2 undergoing uncomplicated appendectomy under general anesthesia

Exclusion Criteria:

* Patient refusal
* drug abuse
* Patient with neurological, psychiatirc or neuromuscular disease
* chronic pain on medicine
* known allergy to the study medicine
* Infection at the site of infiltration

Ages: 14 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Comparison study between Ketamine and Bupivacaine for post operative analgesia | one year
  Analgesia for post -operative Appendectomy operation

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] American Society of Anesthesiologists Task Force on Acute Pain Management. Practice guidelines for acute pain management in the perioperative setting: an updated report by the American Society of Anesthesiologists Task Force on Acute Pain Management. Anesthesiology. 2012 Feb;116(2):248-73. doi: 10.1097/ALN.0b013e31823c1030. No abstract available. PMID 22227789
- [Background] Kehlet H, Holte K. Effect of postoperative analgesia on surgical outcome. Br J Anaesth. 2001 Jul;87(1):62-72. doi: 10.1093/bja/87.1.62. No abstract available. PMID 11460814
- [Background] Barrington JW, Dalury DF, Emerson RH Jr, Hawkins RJ, Joshi GP, Stulberg BN. Improving patient outcomes through advanced pain management techniques in total hip and knee arthroplasty. Am J Orthop (Belle Mead NJ). 2013 Oct;42(10 Suppl):S1-S20. PMID 24911371
- [Background] Baker PN, van der Meulen JH, Lewsey J, Gregg PJ; National Joint Registry for England and Wales. The role of pain and function in determining patient satisfaction after total knee replacement. Data from the National Joint Registry for England and Wales. J Bone Joint Surg Br. 2007 Jul;89(7):893-900. doi: 10.1302/0301-620X.89B7.19091. PMID 17673581